CLINICAL TRIAL: NCT03593538
Title: Effects of Metformin on Mood and Cognition During Nicotine Withdrawal
Brief Title: Effects of Metformin During Nicotine Withdrawal
Acronym: MEP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Pennsylvania Department of Health (Other Government)
Responsible Party: Principal Investigator, Robert Schnoll, Associate Professor, Department of Psychiatry, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 824504
Record Dates: First submitted 2018-06-25; First posted 2018-07-20 (Actual); Results first posted 2021-03-26 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Smoking; HIV-1-infection
MeSH Terms: conditions — Smoking | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low Dose Metformin (Experimental): Days 1-7: Metformin 500 mg per day; Days 8-14: Metformin 500 mg and 1 Placebo capsule per day; Days 15-23: Metformin 500 mg and 2 Placebo capsules per day
  Interventions: Drug: Metformin; Drug: Placebo
- High Dose Metformin (Experimental): Days 1-7: Metformin 500 mg per day; Days 8-14: Metformin 1000 mg per day; Days 15-23: Metformin 1500 mg per day
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Days 1-7: 1 Placebo capsule per day; Days 8-14: 2 Placebo capsules per day; Days 15-23: 3 Placebo capsules per day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Metformin capsule
  Other Names: Glucophage
  Arms: High Dose Metformin; Low Dose Metformin
Drug: Placebo — Sucrose filler in gel capsules
  Other Names: Placebo (for Metformin)
  Arms: Low Dose Metformin; Placebo

SUMMARY:
The purpose of this study is to test the effects of a medication called metformin (Glucophage®) on smoking behavior. This medication is FDA-approved for treatment of type-2 diabetes. It is being used for research purposes in this study. Participants will be randomized to one of 3 treatment groups: low dose of metformin, high dose of metformin, or placebo.

DETAILED DESCRIPTION:
There is a need for novel approaches to optimize smoking cessation treatment to help more smokers quit. Mood disturbance and cognitive deficits during nicotine withdrawal may be important treatment targets given their association with smoking relapse. In addition, factors such as HIV-1 infection may exacerbate abstinence effects on mood and cognitive deficits and thus should be measured and controlled for. The investigators hypothesize that the FDA-approved medication, metformin, will attenuate withdrawal-related mood disturbance and cognitive deficits, controlling for HIV status. Using a well-validated abstinence challenge paradigm, the investigators propose a placebo-controlled double-blind parallel arm study with one between-subjects factor of medication (low dose: 500 mg, high dose: 1500 mg, and placebo). Non-treatment seeking smokers (HIV-: n=54; 18 per group) will complete this 23 day study.

ELIGIBILITY:
Inclusion Criteria

Eligible subjects will be males and females:

1. 18 years of age or older who self-report smoking at least 5 cigarettes (menthol and non-menthol) per day, on average for the past 6 months.
2. HIV status

   1. HIV-infected smokers: diagnosed with HIV infection and exhibiting viral load of less than or equal to 1000 copies/mL and CD4+ counts of greater than or equal to 200 cells/mm3 within 6 months prior to enrollment.
   2. HIV-uninfected smokers: no diagnosis of HIV, either via blood test or self-report.
3. Must not currently be interested in quitting smoking.
4. Women of childbearing potential (based on medical history) must consent to use a medically accepted method of birth control (e.g., condoms and spermicide, oral contraceptive, Depo-Provera injection, contraceptive patch, tubal ligation) or abstain from sexual intercourse during the time they are in the study and using transdermal nicotine.
5. If current or past diagnosis of bipolar disorder, eligible if:

   1. No psychotic features
   2. MADRS: total score less than 8 (past 4 weeks), suicidal item score less than1 (past 4 weeks)
   3. Y-MRS: total score less than 8 (past 4 weeks), irritability, speech content, disruptive or aggressive behavior items score less than 3 (past 4 weeks)
   4. No psychiatric hospitalization or Emergency Room visits for psychiatric issues in the past 6 months
   5. No aggressive or violent acts or behavior in the past 6 months
6. Able to communicate fluently in English.
7. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the combined consent/HIPAA form.

Exclusion Criteria

Smoking Behavior:

1. Current enrollment in a smoking cessation program, or use of other smoking cessation medications in the last month or plans to do either in the next 2 months.
2. Daily use of chewing tobacco, snuff and/or snus, or electronic cigarettes.

Alcohol/Drugs:

1. Self-report current alcohol consumption that exceeds 25 standard drinks/week over the past 6 months. Subjects will be told to limit or avoid the use of alcohol while in the study to avoid any adverse reactions to the study medication.
2. Current untreated and unstable diagnosis of substance dependence (eligible if past use and if receiving treatment and stable for at least 30 days). Current untreated and unstable diagnosis of substance abuse requires Study Physician approval.
3. A positive urine drug screen for cocaine, amphetamines, methamphetamines, PCP, barbiturates and ecstasy (MDMA)at Intake, or any testing session (see Measures and Table 1 for details). Participants believed to have a false-positive result may continue in the study, with investigator approval.

Medical:

1. Females who self-report current pregnancy, planning a pregnancy during the study, or currently breastfeeding/lactating. All female subjects of child-bearing potential shall undergo a urine pregnancy test at the Intake, Baseline, PQ-Testing and 24-H Testing sessions.
2. Current diagnosis of unstable and untreated major depression, as determined by self-report & MINI (eligible if stable for at least 30 days).
3. Current or past diagnosis of psychotic disorder, as determined by self-report or MINI.
4. Suicide risk as indicated by at least one of the following on the MINI/CSSRS (the PI &/or PM [LCSW] will be consulted to assess safety and determine eligibility in cases close to the eligibility cutoffs):

   1. Current suicidal ideation (within 30 days of enrollment)
   2. Two or more lifetime suicide attempts or episodes of suicidal behavior
   3. Any suicide attempt or suicidal behavior within 2 years of enrollment
5. Self-reported kidney and/or liver disease or transplant untreated/unstable or within the past 6 months.
6. Heart/Cardiovascular disease (e.g., angina, coronary heart disease, stroke, etc.) in the past 6 months.
7. Type-1 or type-2 diabetes.
8. Uncontrolled hypertension (BP systolic greater than 159 and/or diastolic greater than 99)*.
9. Liver function tests more than 20% outside of the normal range; Gamma-glutamyl Transpepsidase (GGT) values more than 20% outside of the normal range. If Albumin/Globulin ratios are 20% outside of normal range the abnormal value will be evaluated for clinical significance by the Study Physician and eligibility will determined on a case-by-case basis.
10. Renal disease or renal dysfunction (e.g., serum creatinine levels ≥1.5 mg/dL [males], ≥1.4 mg/dL [females]).
11. A blood glucose level less than 70 mg/dl at any visit.

    * Participants presenting with SBP greater than 159 mmHg and/or DBP greater than 99 mmHg at the Intake visit will be instructed to sit quietly for 10 minutes. Then the participant will have a second blood pressure reading taken after a 10 minute period. If, after the second reading the SBP greater than 159 mmHg and the DBP greater than 99 mmHg, the individual will be ineligible to participate, unless determined otherwise by the Study PI or Study Physician, upon review.

Medication:

1. Current use or recent discontinuation (within the past 14 days) of any of the following medications:

   1. Anti-anxiety or panic disorder medications (e.g., clonazepam, alprazolam).
   2. Anti-psychotic medications as assessed on a case-by-case basis
   3. Glucophage/metformin
   4. Glyburide
   5. Furosemide or digoxin
   6. Nifedipine
   7. Cationic drugs (e.g., amiloride, digoxin, morphine, procainamide, quinidine, quinine, ranitidine, triamterene, trimethoprim, or vancomycin)
2. Participants who report taking prescription opiate-containing medications (Duragesic/fentanyl patches, Percocet, Oxycontin) will require physician approval prior to confirming final eligibility.
3. Current use of any smoking cessation medications (e.g., Chantix/varenicline, Zyban/bupropion, nicotine replacement therapy/gum/patch).
4. For safety reasons, HIV-infected smokers taking dolutegravir (Tivicay) or drugs that contain dolutegravir (e.g., Triumeq) should not take more than 1000 mg of metformin per day. Therefore, individuals taking dolutegravir will be force randomized to either the placebo condition or the low dose condition.

Subjects will be instructed to refrain from using any study prohibited drugs/medications (both recreational and prescription) throughout their participation in the study. After final eligibility is confirmed, subjects who report taking contraindicated medication(s) over the course of the study period may only remain eligible if the Study Physician and/or Principal Investigator determines that the contraindicated medication(s) do/did not impact the study design, data quality, and/or subject safety/welfare. Subjects are permitted to take necessary prescription medications not included within the exclusion list during the study.

General Exclusion:

1. Current, anticipated, or pending enrollment in another research program over the next 2-3 months that could potentially affect subject safety and/or the study data/design as determined by the Principal Investigator and/or Study Physician.
2. Not planning to live in the area for the next two months.
3. Color blindness.
4. Any impairment (physical and/or neurological) including visual or other impairment preventing cognitive task performance.
5. Known allergy to study medication.
6. Planned radiologic studies involving the use of intravascular iodinated contrast materials (e.g., intravenous urogram, intravenous cholangiography, angiography, and computed tomography (CT) scans with intravascular contrast materials) during the course of study participation.
7. Inability to provide informed consent or complete any of the study tasks as determined by the Principal Investigator.
8. Not able to effectively communicate in English (reading, writing, speaking).
9. Missing 3 or more doses during the medication period determined by self-report.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Schnoll, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Center for Interdisciplinary Research on Nicotine Addiction, University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 80 subjects, who signed consent and were deemed eligible to participate, 11 did not attend the Baseline session during which they would begin treatment leaving 69 subjects who started study medication.
Period: Overall Study
Arm/Group | Low Dose Metformin | High Dose Metformin | Placebo
Started | 26 | 21 | 22
Completed | 15 | 15 | 11
Not Completed | 11 | 6 | 11

BASELINE CHARACTERISTICS:
Population: Individuals who started study medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose Metformin | High Dose Metformin | Placebo | Total
Number analyzed (Participants) | 26 | 21 | 22 | 69
Age, Continuous [Mean (Full Range); unit: years] | 49.8 [24 to 67] | 43.1 [20 to 59] | 50.5 [28 to 59] | 47.9 [20 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 7 | 21
  Male | 18 | 15 | 15 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 0 | 4
  Not Hispanic or Latino | 24 | 18 | 22 | 64
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 18 | 17 | 17 | 52
  White | 6 | 2 | 5 | 13
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 1 | 1 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26 | 21 | 22 | 69
Cigarettes per day [Mean (Full Range); unit: cigarettes per day] | 12.6 [4 to 30] | 12.6 [3 to 30] | 16 [6 to 30] | 13.7 [3 to 30]

OUTCOME MEASURES:

1. Primary Outcome: Mood Following 24h of Smoking Abstinence
Description: Self-reported mood on the Positive and Negative Affect Schedule (PANAS), a 20-item Likert-format measure that assesses Positive Affect (PA; 10 items, e.g., enthusiastic, strong) and Negative Affect (NA; 10 items, e.g., distressed, upset). The minimum value for each subscale is 10 and the maximum value is 50. Higher scores indicate greater positive or negative affect.
Time Frame: Day 23
Population: Study Completers
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Low Dose Metformin | High Dose Metformin | Placebo
Number analyzed (Participants) | 15 | 15 | 11
score on a scale
  Positive Affect | 36.5 (2.5) | 33.8 (2.8) | 37.9 (2.6)
  Negative Affect | 14.3 (1.3) | 13.1 (0.9) | 13.9 (1.8)

2. Primary Outcome: Cognitive Function Following 24h of Smoking Abstinence
Description: Composite score of computer-based neurocognitive tasks (N-back Working Memory Task, Stop Signal Task, Hopkins Verbal Learning Test - Revised [HVLT-R]) designed to test working memory and attention. A standardized z-score (mean=0, standard deviation=1) was calculated for the primary outcome for each task and an average was computed from the three z-scores. Higher scores indicated better cognitive performance.
Time Frame: Day 23
Population: Study Completers
Measure: Mean (Standard Error); unit: z-score
Arm/Group | Low Dose Metformin | High Dose Metformin | Placebo
Number analyzed (Participants) | 15 | 15 | 11
z-score | -0.018 (0.17) | 0.159 (0.22) | -0.204 (0.29)

3. Secondary Outcome: Self-reported Smoking Behavior
Description: Cigarettes smoked per day as reported on the Timeline Follow-Back (TLFB). Cigarettes smoked per day is assessed using a "past week" time reference for all time points except the 24-hr testing visit on Day 23, which uses a 24-hr time reference.
Time Frame: Days 7, 14, 21, and 23
Population: Study Completers
Measure: Mean (Standard Error); unit: cigarettes per day
Arm/Group | Low Dose Metformin | High Dose Metformin | Placebo
Number analyzed (Participants) | 15 | 15 | 11
cigarettes per day
  Day 7 | 13.9 (2.2) | 8 (1.1) | 11.2 (1.8)
  Day 14 | 11.8 (1.8) | 8.1 (1.0) | 10.4 (1.8)
  Day 21 | 12.5 (1.7) | 7.4 (0.9) | 10.1 (1.2)
  Day 23 | 0 (0) | 0 (0) | 0 (0)

4. Secondary Outcome: Self-reported Withdrawal Symptoms
Description: The "Minnesota Nicotine Withdrawal Scale - Revised version"(MNWS_R) captures the current state of nicotine withdrawal. The scale assesses eight DSM-IV items of nicotine withdrawal including: dysphoria or depressed mood, insomnia, irritability/frustration/anger, anxiety, decreased heart rate, difficulty concentrating, restlessness, and increased appetite/weight gain. Participants rate the intensity of their symptoms on the following scale: 0 = none, 1 = slight, 2 = mild, 3 = moderate, 4 = severe and a summary score will be calculated. Withdrawal is assessed using a "past week" time reference for all time points except the 24-hr testing visit on Day 23, which uses a 24-hr time reference. The scale ranges from 0 to 32 with higher scores indicating more severe withdrawal symptoms.
Time Frame: Days 7, 14, 21, and 23
Population: Study Completers
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Low Dose Metformin | High Dose Metformin | Placebo
Number analyzed (Participants) | 15 | 15 | 11
score on a scale
  Day 7 | 7.4 (1.3) | 6.3 (0.9) | 7.9 (1.5)
  Day 14 | 7.0 (1.4) | 6.2 (0.8) | 8.3 (2.2)
  Day 21 | 7.8 (1.6) | 5.5 (0.9) | 7.1 (1.7)
  Day 23 | 10.5 (2.1) | 8.7 (1.3) | 11.8 (2.8)

5. Secondary Outcome: Self-reported Craving for Cigarettes
Description: The 10-item brief Questionnaire of Smoking Urges (QSU-B) assesses craving for cigarettes. The QSU-B contains 2 sub-scales (anticipation of reward, relief from negative affect) which are summed to create the total score. Similar to withdrawal symptoms, craving is assessed using a "past week" time reference for all time points except the 24-hr testing visit on Day 23, which will use a 24-hr time reference. Items are rated from 1 (strongly disagree) to 7 (strongly agree) and are summed to create a total score ranging from 10 to 70. Higher scores indicate higher levels of craving.
Time Frame: Days 7, 14, 21, and 23
Population: Study Completers
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Low Dose Metformin | High Dose Metformin | Placebo
Number analyzed (Participants) | 15 | 15 | 11
score on a scale
  Day 7 | 32.9 (4.4) | 26.1 (4.2) | 40.3 (5.8)
  Day 14 | 31.2 (3.6) | 22.3 (3.8) | 38.4 (5.9)
  Day 21 | 28.3 (3.8) | 21.4 (3.3) | 36.7 (5.2)
  Day 23 | 45.2 (5.0) | 39.9 (4.4) | 52.9 (3.8)

6. Secondary Outcome: Subjective Effects of Smoking
Description: The Cigarette Evaluation Scale (CES), developed to assess subjective effects of smoking, is an 11-item Likert-format measure. Questions include items for nausea and dizziness, craving relief, and enjoyment of airway sensations and comprise 3 scales: satisfaction score, psychological relief score, and toxicity score. Each scale is the average of items with a minimum value of 1 and a maximum value of 7. Higher scores indicate more satisfaction, greater psychological relief, and higher subjective toxicity, respectively.
Time Frame: Days 7, 14, 21, and 23
Population: Study Completers
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Low Dose Metformin | High Dose Metformin | Placebo
Number analyzed (Participants) | 15 | 15 | 11
score on a scale
  Satisfaction (Day 7) | 4.7 (0.4) | 3.8 (0.4) | 5.8 (0.4)
  Satisfaction (Day 14) | 5.0 (0.4) | 3.4 (0.5) | 5.2 (0.4)
  Satisfaction (Day 21) | 4.5 (0.4) | 3.6 (0.4) | 5.0 (0.4)
  Satisfaction (Day 23) | 5.1 (0.5) | 3.6 (0.6) | 4.9 (0.6)
  Psychological Relief (Day 7) | 2.7 (0.4) | 2.0 (0.2) | 4.0 (0.6)
  Psychological Relief (Day 14) | 3.0 (0.5) | 2.0 (0.3) | 3.5 (0.5)
  Psychological Relief (Day 21) | 2.8 (0.5) | 1.9 (0.3) | 3.9 (0.6)
  Psychological Relief (Day 23) | 3.2 (0.4) | 2.1 (0.3) | 3.6 (0.5)
  Toxicity (Day 7) | 1.1 (0.06) | 1.4 (0.18) | 1.3 (0.15)
  Toxicity (Day 14) | 1.1 (.08) | 1.6 (0.30) | 1.3 (.15)
  Toxicity (Day 21) | 1.3 (0.11) | 1.2 (0.11) | 1.3 (0.16)
  Toxicity (Day 23) | 2.1 (0.26) | 2.1 (0.26) | 2.6 (0.45)

7. Secondary Outcome: Subjective Sensory Experience of Smoking
Description: The Rose Sensory Questionnaire (SQ), a 9-item Likert-format measure, assesses how much participants liked the cigarette smoked (liking scale) and how high in nicotine the cigarettes appeared to be (strength scale). The questionnaire also includes a diagram of the respiratory tract and asks participants to rate the strength of the cigarette puffs on their tongue, nose, back of mouth and throat, windpipe, and chest. Each scale is the average of items with a minimum value of 1 and a maximum value of 7. Higher scores indicate greater liking and perceived strength, respectively.
Time Frame: Days 7, 14, 21, and 23
Population: Study Completers
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Low Dose Metformin | High Dose Metformin | Placebo
Number analyzed (Participants) | 15 | 15 | 11
score on a scale
  Liking scale (Day 7) | 4.6 (0.33) | 3.8 (0.36) | 5.0 (0.33)
  Liking scale (Day 14) | 4.6 (0.29) | 3.6 (0.44) | 4.8 (0.43)
  Liking scale (Day 21) | 4.4 (0.37) | 3.6 (0.43) | 4.7 (0.29)
  Liking scale (Day 23) | 4.7 (0.36) | 3.7 (0.43) | 4.8 (0.48)
  Strength scale (Day 7) | 3.9 (0.34) | 3.4 (0.45) | 3.9 (0.42)
  Strength scale (Day 14) | 4.0 (0.39) | 2.9 (0.47) | 3.9 (0.39)
  Strength scale (Day 21) | 3.5 (0.43) | 2.9 (0.44) | 3.5 (0.29)
  Strength scale (Day 23) | 4.1 (0.40) | 3.4 (0.51) | 4.0 (0.47)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 30 days
Arm/Group | Low Dose Metformin | High Dose Metformin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/21 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/21 | 0/22
Other Adverse Events (participants affected / at risk) | 12/26 | 11/21 | 14/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose Metformin (N=26) | High Dose Metformin (N=21) | Placebo (N=22)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 1
Headache (General disorders) | 1 | 1 | 3
Heartburn (Gastrointestinal disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 6 | 7 | 5
Increased Sweating (General disorders) | 1 | 1 | 1
Minor Head Injury (General disorders) | 1 | 0 | 0
Mouth Sores (General disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 0
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-17): https://cdn.clinicaltrials.gov/large-docs/38/NCT03593538/Prot_SAP_000.pdf
  • Informed Consent Form (2020-11-09): https://cdn.clinicaltrials.gov/large-docs/38/NCT03593538/ICF_001.pdf